CLINICAL TRIAL: NCT02319902
Title: The Effects of Using Heated Humidified Carbon Dioxide Gas on Post Operative Pain Scores, Nausea and Analgesic Requirements in Patients Undergoing Gynaecological Laparoscopy: a Randomised Controlled Trial.
Brief Title: Standard Carbon Dioxide Gas Versus Heated Humidified Gas in Gynaecological Laparoscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fevzi Shakir (Other)
Responsible Party: Sponsor-Investigator, Fevzi Shakir, Senior Clinical Research Fellow in Advanced Gynaecological Laparoscopic Surgery, Royal Surrey County Hospital NHS Foundation Trust
Organization: Royal Surrey County Hospital NHS Foundation Trust (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14SURN0015
Record Dates: First submitted 2014-12-14; First posted 2014-12-18 (Estimated); Last update posted 2014-12-18 (Estimated); Status verified 2014-12

CONDITIONS: Heated Humidified Carbon Dioxide in Gynaecological Laparoscopic Surgery

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard cold carbon dioxide gas (Placebo Comparator): Standard cold carbon dioxide gas
  Interventions: Device: Standard cold carbon dioxide gas
- Heated humidified carbon dioxide gas (Active Comparator): Heated humidified carbon dioxide gas
  Interventions: Device: Heated humidified carbon dioxide gas

INTERVENTIONS:
Device: Standard cold carbon dioxide gas — Use of standard cold carbon dioxide gas in laparoscopic gynaecological surgery.
  Arms: Standard cold carbon dioxide gas
Device: Heated humidified carbon dioxide gas — Use of the Fischer and Paykel heated humidification system for laparoscopic gynaecological surgery.
  Arms: Heated humidified carbon dioxide gas

SUMMARY:
To establish if heated humidified carbon dioxide gas improves pain scores as well as nausea and analgesic requirements in post operative patients compared to standard cold carbon dioxide.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age
* Patients planned to undergo laparoscopy for minor procedures such as endometriosis, adhesions, ovarian cystectomies, bilateral salpingoophorectomy, tubal ligation and sterilisation will be invited to participate in the trial.
* Capacity to consent

Exclusion Criteria:

* Patients unable to speak English
* Patients unable to give consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2014-12; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Shoulder tip pain | 8 hours
  Shoulder tip pain recorded as a visual analogue scale from 1-10, 8 hours post surgery compared to baseline

SECONDARY OUTCOMES:
General abdominal pain, nausea, vomiting and analgesia requirements | 8 hours
  General abdominal pain, nausea, vomiting and analgesia requirements 8 hours post surgery compared to baseline
Shoulder tip pain, general abdominal pain, nausea, vomiting. | 7 days
  Shoulder tip pain, general abdominal pain, nausea, vomiting over a 7 day period compared to baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Surrey County Hospital NHS Trust, Guildford, Surrey, United Kingdom